CLINICAL TRIAL: NCT04873544
Title: Enhanced Recovery After Surgery Protocols in Total Knee Arthroplasty Via Midvastus Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY20170418-02
Record Dates: First submitted 2021-04-30; First posted 2021-05-05 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2020-07

CONDITIONS: ERAS; Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Common protocols for TKA (Experimental): Common protocols for TKA
  Interventions: Procedure: ERAS protocols for TKA

INTERVENTIONS:
Procedure: ERAS protocols for TKA — ERAS protocols for TKA

SUMMARY:
The study aimed to investigate the impact of enhanced recovery after surgery (ERAS) protocols on the clinical effect of total knee arthroplasty (TKA) via the midvastus approach

DETAILED DESCRIPTION:
In this study, a randomized controlled study was conducted to further investigate the impact of ERAS protocols in the clinical efficacy of TKA with the midvastus approach. The ERAS protocols were adopted for the ERAS group and consisted of pure juice drinking 2 hours before the surgery, optimization of the preoperative anesthesia plan, phased use of tourniquets, and the use of tranexamic acid as well as a drug cocktail. The operative time, first postoperative walking time, first straight leg elevation time, postoperative hospitalization time, visual analogue scale score (VAS score), New York Hospital of Special Surgery knee score (HSS score), Knee Society Score (KSS score), and knee range of motion were used to assess the clinical effects in the two groups. All the included patients were followed up for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral primary knee osteoarthritis
* Varus, valgus, and flexion contracture deformity of the knee joint < 10°
* The range of motion of the knee joint was > 80°
* Body mass index (BMI) < 30
* No previous history of knee surgery on the affected side .Agreed to participate in the trial.

Exclusion Criteria:

* Rheumatoid arthritis
* Extra-knee deformity
* Simultaneous bilateral knee arthroplasty
* Severe dysfunction of the liver, kidney, and blood system
* Severe cardiovascular diseases
* Gastrointestinal ulcer .Other medical conditions like nausea, vomiting, snoring, and allergy to related analgesic drugs.

Ages: 56 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
the postoperative hospitalization time | 12 months
  the postoperative hospitalization time

SECONDARY OUTCOMES:
the operative time | 2 hours
  the operative time
first postoperative walking time | 1 day
  first postoperative walking time
first straight leg elevation time | 1 day
  first straight leg elevation time
visual analogue scale score (VAS score) | 12 months
  VAS score (0-10 scores) is for pain: 0 represent no pain, 1-3 represent mild pain, 4-6 represent moderate pain, 7-10 represent severe pain.
New York Hospital of Special Surgery knee score (HSS score) | 12 months
  HSS score (0-100 scores) is for knee function: 85-100 represent excellent, 70-84 represent good, 60-69 represent fair, 0-59 represent bad.
Knee Society Score (KSS score) | 12 months
  KSS score (0-100 scores) is for knee function: 85-100 represent excellent, 70-84 represent good, 60-69 represent fair, 0-59 represent bad.
knee range of motion | 12 months
  knee range of motion

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing first hospital, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Wei B, Tang C, Li X, Lin R, Han L, Zheng S, Xu Y, Yao Q, Wang L. Enhanced recovery after surgery protocols in total knee arthroplasty via midvastus approach: a randomized controlled trial. BMC Musculoskelet Disord. 2021 Oct 8;22(1):856. doi: 10.1186/s12891-021-04731-6. PMID 34625057